Comparison of the Effects of Personal Versus Hospital-Provided Dolls on Preoperative Anxiety and Postoperative Delirium in Preschool Children

**Document Type:** Study Protocol **Ethics Committee Approval Date:** 14 January 2026

## **Brief Description**

The goal of this study is to evaluate the effects of personal versus hospital-provided dolls on preoperative anxiety and postoperative delirium in preschool children aged 3–7 years undergoing elective adenoidectomy and/or tonsillectomy.

### **Study Design**

This study is designed as a prospective observational study.

### **Study Population**

Female children aged 3–7 years scheduled for elective adenoidectomy and/or tonsillectomy under general anesthesia.

## **Eligibility Criteria**

<u>Inclusion Criteria:</u> Female children aged 3–7 years• Scheduled for elective adenoidectomy and/or tonsillectomy under general anesthesia• Able to communicate verbally• ASA physical status I or II, according to the American Society of Anesthesiologists classification• Written informed consent obtained from a parent or legal guardian <u>Exclusion Criteria:</u> Presence of psychiatric, neurological, or developmental disorders• Presence of chronic pain or ongoing medical treatment that may affect anxiety levels• Refusal to participate despite repeated encouragement by the investigators• Use of additional anxiety-reducing methods or medications outside the study protocol prior to intervention• Previous surgical experience

#### **Study Procedures**

Eligible participants will be observed during the routine perioperative period and categorized into one of three groups based on doll use: hospital-provided doll, personal doll, or no doll. Preoperative anxiety levels will be assessed at predefined time points using standardized anxiety scales. Serum cortisol levels will be measured from an additional blood sample obtained during routine intravenous cannulation without requiring any extra invasive procedures. Postoperative emergence delirium will be evaluated in the post-anesthesia care unit using a validated pediatric delirium scale.

#### **Outcome Measures**

Preoperative anxiety will be assessed using the Modified Yale Preoperative Anxiety Scale (m-YPAS) and Visual Analog Scale for Anxiety (VAS-A). Postoperative emergence delirium will be assessed using the Pediatric Anesthesia Emergence Delirium (PAED) scale.

#### **Timing of Assessments**

Preoperative assessments: waiting area, before transfer, during transfer, before anesthesia induction.

Postoperative assessments: immediately after extubation, upon admission to the post-anesthesia care unit, and 30 minutes after admission.

# **Statistical Analysis**

Descriptive statistics will be used. Between-group comparisons will be performed using appropriate parametric or non-parametric tests based on data distribution. A p-value < 0.05 will be considered significant.

## **Ethics**

The study will be conducted in accordance with the Declaration of Helsinki. Ethics committee approval and written informed consent from parents/legal guardians will be obtained.